CLINICAL TRIAL: NCT07164287
Title: Retrospective Observational Study of Intensity Effects in Psychedelic-assisted Treatment
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Louise Penzenstadler, Principal investigator, University Hospital, Geneva
Other Study IDs: ID 2022-02015
Record Dates: First submitted 2025-08-22; First posted 2025-09-10 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder (MDD); Anxiety Disorders; Substance Use Disorder (SUD); PTSD - Post Traumatic Stress Disorder
Keywords: psychedelic; LSD; psilocybin
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders; Substance-Related Disorders; Combat Disorders | interventions — Lysergic Acid Diethylamide; Psilocybin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Lysergic Acid Diethylamide (LSD) or psilocybin — Psychedelic-assisted psychotherapy with LSD or psilocybin as a part of a clinical routine in our department

SUMMARY:
This retrospective observational study examines the effects of psychedelic-assisted psychotherapy (PAP) with lysergic acid diethylamide (LSD) or psilocybin in patients with treatment-resistant depressive, anxiety, or addictive disorders.

Data will be analyzed from patients treated at the University Hospitals of Geneva between June 2020 and April 2025 who obtained individual authorizations from the Swiss Federal Office of Public Health for use of LSD or psilocybin under compassionate use criteria.

The main objective is to assess the effects of psychedelic-assisted psychotherapy with LSD or psilocybin on changes in depressive symptoms, anxiety symptoms. Secondary objectives include evaluating the association between psychedelic session intensity and the administered dose of LSD or psilocybin, changes in depressive symptoms, anxiety symptoms, and problematic substance use, as well as their association with intensity effects. Additionally physiological effects during session will be assessed.

All data are retrospectively collected from clinical records with prior patient consent.

This study aims to generate evidence on the feasibility, safety, and therapeutic potential of PAP in real-world clinical practice.

DETAILED DESCRIPTION:
The overall project is a retrospective observational study evaluating the effects of psychedelic-assisted psychotherapy (PAP) with LSD or psilocybin in treatment-resistant depressive, anxiety, and addictive disorders. Data from 200 patients treated at Geneva University Hospitals will be included, with the primary aim of assessing relationships between psychedelic dose, subjective intensity of experience, and clinical outcomes.

Subset Analysis: Cardiovascular Outcomes In addition to the main objectives, a subset analysis will be conducted to evaluate cardiovascular effects of LSD and psilocybin. Routinely collected data from 30 patients with treatment-resistant depression or anxiety disorders will be included.

Population: 30 patients who underwent their first psychedelic session (LSD 100-200 µg or psilocybin 15-25 mg).

Measurements: Heart rate and self-rated anxiety (visual analogue scale) recorded at seven time points between 30 and 300 minutes post-administration on the treatment day.

A further subset analysis investigated the role of early maladaptive schemas (EMS) in psychedelic-assisted psychotherapy.

Populations: 192 patients who routinely completed the Young Schema Questionnaire - Rasch version (YSQ-R) before treatment were included; of these, 97 initiated PAP with LSD or psilocybin and 74 contributed longitudinal outcomes.

Measurements: Baseline EMS profiles (YSQ-R) measured at Baseline (screening or preparation visit, before first psychedelic session), immediately after each psychedelic session (sessions 1-3, up to 9 months) and 1 month after each psychedelic session (sessions 1-3, up to 12 months after baseline).

ELIGIBILITY:
Inclusion Criteria:

* Patients treated in the compassionate PAP program at Geneva University Hospitals between June 2020 and April 2025.
* Diagnosis of depressive, anxiety, or addictive disorder resistant to standard treatments.
* General consent for use of routinely collected clinical data.
* Federal Office of Public Health authorization for PAP.

Exclusion Criteria:

* psychotic disorder
* bipolar disorder
* high suicidal risk
* severe cardiovascular disease
* severe liver disease
* neurological disease of the central nervous system
* pregnancy
* breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with treatment-resistant depressive, anxiety, or addictive disorders who received psychedelic-assisted psychotherapy under compassionate use authorization treated in the psychedelic-assisted psychotherapy program at Addiction Division, Department of Psychiatry, Geneva University Hospital, Switzerland.
Sampling Method: Non-Probability Sample
Enrollment: 376 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Self-reported depressive symptoms (BDI-II) | Baseline and 1 month after each psychedelic treatment session (sessions 1-3, up to 12 months)
  Beck Depression Inventory-II, total scores ranging from 0 to 63, higher scores indicating higher depressive symptoms
Self-reported symptoms of anxiety (STAI) | Baseline and 1 month after each psychedelic treatment session (sessions 1-3, up to 12 months)
  State-Trait Anxiety Inventory, total scores ranging from 20 to 80, higher scores indicating higher anxiety

SECONDARY OUTCOMES:
Self-reported intensity of mystical experience | the day of treatment administration
  Assessed with the self-report Mystical experience Questionnaire (MEQ-30) with total man score ranging from 0 to 5, with higher scores indicating higher intensity of mystical experience
heart rate | day of treatment administration
  beats per minute
Self-rated anxiety | day of treatment administration
  Self-rated anxiety using a 0-100 visual analogue scale (VAS), with higher scores indicating higher anxiety
Young Schema Questionnaire - Rasch version | Baseline (screening or preparation visit, before first psychedelic session), immediately after each psychedelic session (sessions 1-3, up to 9 months) and 1 month after each psychedelic session (sessions 1-3, up to 12 months after baseline)
  116-item self-report questionnaire assessing 20 early maladaptive schemas. Items are rated on a 6-point Likert scale (1 = completely untrue of me, 6 = describes me perfectly). Higher scores indicate greater schema intensity; schema-specific and overall mean scores can be derived.

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided